CLINICAL TRIAL: NCT06169098
Title: Changes in Skin Surface Temperature of the Lumbar Region During Auricular Acupressure at Kidney Point on Healthy Volunteers
Brief Title: Changes in Lumbar Region Temperature During Auricular Acupressure at Kidney Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 699/HDDD-DHYD
Record Dates: First submitted 2023-11-28; First posted 2023-12-13 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AA-SA (Experimental): Order: auricular acupressure on the left ear, auricular acupressure on the right ear, sham auricular acupressure on the left ear.
  There will be a 30-minute break between each stage.
  Interventions: Procedure: Auricular acupressure on the left ear; Procedure: Auricular acupressure on the right ear; Procedure: Sham auricular acupressure
- SA-AA (Experimental): Order: sham auricular acupressure on the left ear, auricular acupressure on the right ear, auricular acupressure on the left ear.
  There will be a 30-minute break between each stage.
  Interventions: Procedure: Auricular acupressure on the left ear; Procedure: Auricular acupressure on the right ear; Procedure: Sham auricular acupressure

INTERVENTIONS:
Procedure: Auricular acupressure on the left ear — Auricular acupressure is applied at the Kidney point on the left ear using a tape with a Vaccaria seed (2mm in diameter). After placement on this acupoint, apply consistent moderate pressure for 5 minutes.
Procedure: Auricular acupressure on the right ear — Auricular acupressure is applied at the Kidney point on the right ear using a tape with a Vaccaria seed (2mm in diameter). After placement on this acupoint, apply consistent moderate pressure for 5 minutes.
Procedure: Sham auricular acupressure — Sham auricular acupressure is applied at Kidney point on the left ear using a tape without any seed. After placement on this acupoint, apply consistent moderate pressure for 5 minutes.

SUMMARY:
In Traditional Medicine, auricular acupressure (AA) is one of the non-pharmacological treatment methods commonly utilized due to its safety and convenience. AA involves the application of a taped seed of Vaccaria (with a diameter of 2mm) on specific ear acupoints to manage various disorders. Among these, chronic lower back pain is prevalent. According to Traditional Medicine, the Kidney point is selected for this condition due to the belief that "The lumbar region is the house of the Kidneys". However, evidence supporting this correlation is still lacking. In this study, the aim is to assess the relationship between the Kidney point and the lumbar region by monitoring changes in skin temperature through the application of AA on this acupoint.

DETAILED DESCRIPTION:
Healthy volunteers meeting all selection criteria and not violating exclusion criteria will be recruited for the study.

Before commencement, participants will acclimate to the environment for 15 minutes, allowing stabilization of blood pressure, heart rate, respiratory rate, and body temperature. The room will be enclosed and shielded, ensuring no direct sunlight or other radiation sources enter. Room temperature, pressure, humidity, and ventilation will be consistently maintained throughout the study.

The participants will be randomly divided into two groups: one receiving auricular acupressure (AA) first followed by sham auricular acupressure (SA) (AA-SA group), while the other group will receive SA first followed by AA (SA-AA group).

Blood pressure, heart rate, respiratory rate, body temperature, lumbar region temperature, and side effects of auricular therapies will be continuously monitored.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 23 kg/m2.
* Demonstrates alertness and cooperativeness.
* Vital signs within normal limits.
* Voluntary informed consent.

Exclusion Criteria:

* Anxiety, depression, or stress based on the Depression Anxiety and Stress Scales 21 (DASS-21).
* Presence of disorders or use of medications affecting body temperature.
* Received any form of heat therapy for the lower back within the past week (e.g., acupuncture, heat pads, patches, massage).
* Applied chemical or pharmaceutical products to the skin area under investigation prior to the study.
* Current disorders or pathologies in the lumbar region.
* Engaged in nighttime activities or experienced insomnia the night before the research day.
* Participated in sports activities within 2 hours before the study.
* Used stimulants within 24 hours prior.
* History of alcohol or substance addiction.
* History of hypersensitivity reactions to any form of acupuncture.
* Existing injuries or lesions at acupoints and areas investigated in this study.
* Women currently menstruating, pregnant, or breastfeeding.
* Prior experience with auricular therapies.
* Currently participating in other intervention studies.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Change in temperature of the left lumbar region | During procedure
  The temperature of the lumbar region is recorded using an infrared thermal imaging camera. The unit is degrees Celsius (°C).
Change in temperature of the right lumbar region | During procedure
  The temperature of the lumbar region is recorded using an infrared thermal imaging camera. The unit is degrees Celsius (°C).

SECONDARY OUTCOMES:
The proportion of auricular acupuncture side effects | During procedure

OTHER OUTCOMES:
Change in body temperature | During procedure
  Body temperature is measured in the armpit using a digital thermometer. The unit is degrees Celsius (°C).
Change in heart rate | During procedure
  The unit is beat per minute (bpm).
Change in respiratory rate | During procedure
  The unit is breath per minute (bpm).
Change in blood pressure | During procedure
  Blood pressure is measured on the arm using an electronic blood pressure monitor, including systolic and diastolic blood pressure. The unit is mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Moura CC, Chaves ECL, Chianca TCM, Ruginsk SG, Nogueira DA, Souza VHS, Iunes DH. Contribution of Chinese and French ear acupuncture for the management of chronic back pain: A randomised controlled trial. J Clin Nurs. 2019 Nov;28(21-22):3796-3806. doi: 10.1111/jocn.14983. Epub 2019 Aug 9. PMID 31237981
- [Background] Guan L, Li G, Yang Y, Deng X, Cai P. Infrared thermography and meridian-effect evidence and explanation in Bell's palsy patients treated by moxibustion at the Hegu (LI4) acupoint: Overall regulation or a specific target? Neural Regen Res. 2012 Mar 25;7(9):680-5. doi: 10.3969/j.issn.1673-5374.2012.09.007. PMID 25745463
- [Background] Fan AY, Miller DW, Bolash B, Bauer M, McDonald J, Faggert S, He H, Li YM, Matecki A, Camardella L, Koppelman MH, Stone JAM, Meade L, Pang J. Acupuncture's Role in Solving the Opioid Epidemic: Evidence, Cost-Effectiveness, and Care Availability for Acupuncture as a Primary, Non-Pharmacologic Method for Pain Relief and Management-White Paper 2017. J Integr Med. 2017 Nov;15(6):411-425. doi: 10.1016/S2095-4964(17)60378-9. PMID 29103410
- [Background] Hou PW, Hsu HC, Lin YW, Tang NY, Cheng CY, Hsieh CL. The History, Mechanism, and Clinical Application of Auricular Therapy in Traditional Chinese Medicine. Evid Based Complement Alternat Med. 2015;2015:495684. doi: 10.1155/2015/495684. Epub 2015 Dec 28. PMID 26823672
- [Background] Moura CC, Iunes DH, Ruginsk SG, Souza VHS, Assis BB, Chaves ECL. Action of ear acupuncture in people with chronic pain in the spinal column: a randomized clinical trial1. Rev Lat Am Enfermagem. 2018 Sep 3;26:e3050. doi: 10.1590/1518-8345.2678.3050. PMID 30183875
- [Background] Tan JY, Molassiotis A, Wang T, Suen LK. Adverse events of auricular therapy: a systematic review. Evid Based Complement Alternat Med. 2014;2014:506758. doi: 10.1155/2014/506758. Epub 2014 Nov 10. PMID 25435890
- [Background] Gao XY, Zhang SP, Zhu B, Zhang HQ. Investigation of specificity of auricular acupuncture points in regulation of autonomic function in anesthetized rats. Auton Neurosci. 2008 Feb 29;138(1-2):50-6. doi: 10.1016/j.autneu.2007.10.003. PMID 18068545
- [Background] He W, Wang X, Shi H, Shang H, Li L, Jing X, Zhu B. Auricular acupuncture and vagal regulation. Evid Based Complement Alternat Med. 2012;2012:786839. doi: 10.1155/2012/786839. Epub 2012 Nov 27. PMID 23304215
- [Background] Morrison SF, Nakamura K. Central Mechanisms for Thermoregulation. Annu Rev Physiol. 2019 Feb 10;81:285-308. doi: 10.1146/annurev-physiol-020518-114546. Epub 2018 Sep 26. PMID 30256726